CLINICAL TRIAL: NCT03226548
Title: An Experimental Investigation Into the Impact of Socioeconomic Context on Biological Markers of Aging, Health and Mortality
Brief Title: Effect of EITC on Biological Markers of Aging, Health and Mortality
Acronym: PaycheckPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: MDRC (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAQ9663 (ADD-ON); R01AG054466 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Poverty; Tax Policy
Keywords: Earned Income Tax Credit (EITC); Tax Credit; Paycheck Plus

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Paycheck Plus: Participants will receive four times the standard Earned Income Tax Credit after filing their annual taxes
  Interventions: Other: Paycheck Plus
- Control (No Intervention): Control participants will receive the standard Earned Income Tax Credit after filing their annual taxes

INTERVENTIONS:
Other: Paycheck Plus — A four-fold increase in the Earned Income Tax Credit
  Arms: Experimental

SUMMARY:
Paycheck Plus (PP) is a randomized controlled experiment (RCT) that explores the health and longevity effects associated with increasing the Earned Income Tax Credit (EITC). EITC is a national program that provides tax credits to low-income, disproportionately minority workers who file taxes. EITC is politically popular, having received bipartisan support. The EITC, along with state supplemental programs, have 7 million American families out of poverty. The investigators' preliminary data analyses show that the EITC has had large population health impacts, reversing declines in self rated health and survival among the poorest Americans.

DETAILED DESCRIPTION:
Poverty disproportionately impacts minority and rural populations and is very strongly correlated with poor health over the life cycle, and has been hypothesized to lead to a shorter, less healthy aging process. Poverty is associated with a greater burden of disease than smoking and obesity combined and accounts for the bulk of health disparities by race. It is widely believed that an antipoverty policy, such as Earned Income Tax Credit (EITC), could improve healthy aging among working-age low-income adults over the life cycle. It does so by increasing material hardship and psychological stress, two risk factors that are strongly correlated with biological markers of premature aging (e.g., shorter telomeres, higher cholesterol levels, and higher blood pressure).

ELIGIBILITY:
Inclusion Criteria:

1. a US resident
2. Filed taxes
3. Earned <$30,000 in the previous year
4. Aged 21-64
5. Have a Social Security number

Exclusion Criteria:

1. Eligible for Supplemental Security Income or Social Security Disability Insurance
2. Married
3. Have dependent children

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1350 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Score on the Patient Health Questionnaire-9 (PHQ-9) | 4 Years
  Depression will be measured using the subject's score on the PHQ-9.
EuroQol 5D5L | 4 years
  Health-related quality of life

SECONDARY OUTCOMES:
Mean Body Mass Index (BMI) | 2 Years
  A measure of obesity
Telomere length | 4 years
  Telomere length is a measure of biological age
Mortality | 4 years
  We will link records to National Death Index for future study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Muennig, MD, Principal Investigator — Columbia University
Locations (1):
- Westat, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy we cannot share our data